CLINICAL TRIAL: NCT01588717
Title: A Pilot Study to Measure and Treat Antidepressant-Induced Excessive Sweating With Glycopyrrolate (AIDES-G)
Brief Title: Excessive Sweating Caused by Antidepressants: Measurement and Treatment With Glycopyrrolate (AIDES-G)
Acronym: AIDES-G
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIDES-G
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Hyperhydrosis; Depression
Keywords: Hyperhydrosis; Excessive Sweating; Sweating; Depression; Antidepressant
MeSH Terms: conditions — Hyperhidrosis; Depression | interventions — Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- glycopyrrolate (Experimental): glycopyrrolate 2 to 6 mg/day
  Interventions: Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Glycopyrrolate — glycopyrrolate 2 to 6mg/day
  Other Names: Cuvposa®; Robinul®; Robinul® Forte

SUMMARY:
The study consists of measurement of antidepressant-induced excessive sweating and its treatment with an experimental medication, glycopyrrolate (approved to treat ulcers), which will be added to the antidepressant. This is an open-label study (no placebo group or concealment of the nature of the treatment) that will last 8 weeks, including two weeks of baseline measurement without treatment with the study medication followed by six weeks of treatment with the study medication. The study is pilot study by Dr. Rajnish Mago that is based on the hypothesis that glycopyrrolate will be effective in reducing the severity of excessive sweating caused by antidepressant treatment, and will have minimal side-effects.

DETAILED DESCRIPTION:
Sweating is a common and bothersome adverse effect of treatment with antidepressants. Tricyclics and selective serotonin reuptake inhibitors (SSRIs) have both been clearly shown to cause sweating. Increased sweating has been reported with venlafaxine (Pierre and Guze, 2000) and bupropion (Feighner et al. 1984) as well. It is unclear to what extent tolerance develops to antidepressant-induced sweating. It may continue to be a problem even after 6 or more months on the antidepressant (e.g., Mavissakalian et al., 2002).

The prevalence of sweating with SSRIs is estimated to be between 7% and 19% depending on the drug (Ashton & Weinstein 2002). According to the Physician's Desk Reference, excessive sweating occurs in 3-11% patients in clinical trials of SSRIs. Considering the fairly high prevalence of excessive sweating during antidepressant use and its consequences of patient distress and treatment noncompliance, it is important that more intensive efforts be made to understand the phenomenon and to systematically study potential treatments for it.

The mechanism of antidepressant-induced sweating has not been clearly elucidated and there is no generally accepted treatment for it. Initially, a reduction in the dose may be attempted to resolve antidepressant-induced sweating. However, a reduction of dose may not always be helpful (Leeman, 1990; Ashton & Weinstein 2002) as it has been noted that the presence of sweating is not a clear dose-related symptom. As well, reducing the dose of the antidepressant may lead to a worsening of depression and therefore be an unrealistic alternative.

Antiadrenergic drugs like clonidine and terazosin (Feder, 1995; Mago and Monti, 2007; Mago et al., 2009) may be effective for the treatment of antidepressant-induced excessive sweating because the nervous system control of sweating is initially mediated by adrenergic receptors. However, antiadrenergic treatment may be associated with a decrease in blood pressure in some patients, which may lead to dizziness, especially on standing up. Also, the improvement in excessive sweating may not be complete.

Therefore, additional approaches are needed. Sweat glands are innervated by nerve fibers that release acetylcholine. Anticholinergic medications could be used as a potential treatment for the excessive sweating. In case reports, the anticholinergic drug benztropine has been successfully used to treat antidepressant-induced excessive sweating (Garber and Gregory, 1997; Feder and Guze, 2000). However, this has not been confirmed in a clinical trial. Also, benztropine readily crosses the blood-brain barrier; therefore, in addition to its desired effect peripherally on the sweat glands, it tends to cause cognitive side effects through its central effects.

Glycopyrrolate is an anticholinergic medication that is preferred for a variety of clinical uses because it does not cross the blood-brain barrier to a great extent. It has been used for many years by anesthesiologists to dry secretions during surgical procedures. In a case series based on chart review (Tran et al., 2009), it was found to be effective for antidepressant-induced excessive sweating.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Presence of excessive sweating by self-report
3. Within 2 months of initiation of an antidepressant or increase in the dose, there was a clear and substantial increase in sweating not explained by undue external warmth, exercise, or other reason. If treatment with the antidepressant was interrupted, did not persist for more than 6 weeks during that interruption
4. Treatment with the antidepressant is deemed to be clinically necessary due to substantial benefit from the antidepressant that is causing the excessive sweating, and failure to respond to or tolerate an alternative antidepressant
5. Decrease in dose of the antidepressant is either not clinically viable due to the benefit obtained at the current dose OR decrease in dose of the antidepressant has been tried but was not effective.
6. Excessive sweating has persisted for at least 4 weeks prior to baseline assessment
7. The excessive sweating is rated by the patient as at least moderately bothersome.
8. Episodes of excessive sweating occur at least twice a week for last 4 weeks
9. Use of effective contraception (e.g., sterilization, oral contraceptives, condom with spermicide, etc)

Exclusion Criteria:

1. Presence of another known disease that could potentially cause excessive sweating
2. Failure to respond in the past to anticholinergic treatment for excessive sweating
3. Previous allergic reaction to glycopyrrolate
4. Narrow angle glaucoma
5. Significant cardiac disease including cardiac or heart block
6. Patients with known hot-flashes or who are menopausal
7. History of urinary retention
8. History of seizures
9. Pregnancy or breastfeeding
10. Other significant medical illness or laboratory abnormalities that, in the judgment of the PI, would increase risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression- Improvement scores | 9 weeks per subject
  The main comparison will be the end-of-study mean v. the baseline mean

SECONDARY OUTCOMES:
change in mean of patient rated severity of sweating for each week, and change in mean skin conductance for each week | 9 weeks per subject

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mago, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States